CLINICAL TRIAL: NCT04709757
Title: Intermittent Dosing of Spinal Cord Stimulation as Alternate Paradigm to Continuous 10kHz Frequency Therapy (HF10 Therapy)
Brief Title: Comparison of Continuous and Burst High Frequency Spinal Cord Stimulation Paradigms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Intermittent paradigm replaced with change in frequency and amplitude. The updated protocol is NCT04909138
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Lubenow, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20121301
Record Dates: First submitted 2021-01-06; First posted 2021-01-14 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain; CRPS; Peripheral Neuropathy
Keywords: Chronic pain; Spinal cord stimulation; CRPS
MeSH Terms: conditions — Peripheral Nervous System Diseases; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive 1) Intermittent Dosing Therapy 30 seconds ON 90 seconds OFF or 2) Intermittent Dosing Therapy 30 seconds ON and 360 seconds OFF
  Patients will be seen and evaluated prior to randomization, and thereafter at 2, 4 and 6 weeks. At the 6-week time period, patients will be crossed over to the other study arm and thereafter evaluated at 2, 4 and 6 weeks.
Who Masked: Participant
Masking Description: Participants will not know to which treatment they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intermittent Dosing HF10 30/90 (Active Comparator): Stimulation delivered at 30 seconds ON and 120 seconds OFF through patient's existing spinal cord stimulator.
  Interventions: Device: Intermittent Dosing HF10 30/90
- Intermittent Dosing HF10 30/360 (Active Comparator): Stimulation delivered at 30 seconds ON and 360 seconds OFF through patient's existing spinal cord stimulator.
  Interventions: Device: Intermittent Dosing HF10 30/360

INTERVENTIONS:
Device: Intermittent Dosing HF10 30/90 — 10kHz frequency spinal cord stimulation delivered at 30 seconds ON and 120 seconds OFF
  Arms: Intermittent Dosing HF10 30/90
Device: Intermittent Dosing HF10 30/360 — 10kHz frequency spinal cord stimulation delivered at 30 seconds ON and 360 seconds OFF
  Arms: Intermittent Dosing HF10 30/360

SUMMARY:
Spinal cord stimulation (SCS) delivered at 10kHz frequency (HF10 Therapy) has demonstrated superiority to traditional SCS for leg and back pain. Intermittent dosing (ID) refers to the cycling of stimulation, in which there is a designated time period of stimulation being active (ON) and inactive (OFF). Previous studies have demonstrated the safe and effective use of intermittent dosing. However, there still remains a paucity of clinical data on the use of intermittent dosing and which doses (i.e. on/off cycle time periods) are most effective. Furthermore, no previous studies have utilized HF10 therapy when evaluating intermittent dosing.

Patients with chronic back and/or leg pain who have undergone permanent spinal cord stimulator implantation delivered by the Nevro Omnia Neurostimulation System and who are reporting decreased efficacy of continuous HF10 therapy will be randomized into one of two treatments: 1) Intermittent Dosing therapy at 30 seconds ON, 90 seconds OFF 2)Intermittent Dosing therapy at 30 seconds ON, 360 seconds OFF.

After randomization, each consented subject will present to clinic at which time will first be seen by a team of investigators, sub-investigators, and/or study staff. After evaluation and collection of baseline data, a clinical specialist for the Nevro Omnia Neurostimulation system will program the subject's SCS system according to the treatment group to which they have been randomized, under direct physician supervision

Patient's will be seen and evaluated prior to randomization, and thereafter at 2, 4 and 6 weeks. At the 6-week time period, patients will be crossed over to the other study arm and thereafter evaluated at 2, 4 and 6 weeks.

As our primary endpoint, we hypothesize that ID HF10 therapy will provide non-inferior pain relief as measured by VAS scores when compared to continuous HF10 therapy. Other endpoints include: charging frequency, EQ-5D scores of wellbeing; PROMIS score for physical function, pain interference, sleep disturbance, and emotional distress; chronic pain acceptance questionnaire 8 (CPAQ-8), patient satisfaction scores, and patient global impression of change

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) delivered at 10kHz frequency (HF10 Therapy) has demonstrated superiority to traditional SCS for leg and back pain. This mode of stimulation entails delivery of a greater charge per second compared to traditional tonic spinal cord stimulation and corresponding implications for battery usage. Although not yet studied in novel modes of SCS such as HF10 and Burst3 due to their relative infancy, the possibility of decreased pain relief over time very much exists. This has been well-documented with the use of tonic spinal cord stimulation. Furthermore, the most common cause of spinal cord stimulator explant remains the lack or loss of efficacy. In order to mitigate the potential for waning pain relief over time and downstream consequences of increased charge burden, other paradigms of stimulation within the framework of HF10 therapy must be evaluated.

Intermittent dosing (ID) refers to the cycling of stimulation, in which there is a designated time period of stimulation being active (ON) and inactive (OFF). Previous studies have demonstrated the safe and effective use of intermittent dosing. In 2020, Deer et al. reported the efficacy of intermittent dosing of Burst stimulation with settings ranging from 30 seconds ON and 90 seconds OFF, to 30 seconds ON and 360 seconds OFF. In this 50 subject study, 45.8% of patients preferred stimulation with 30 seconds ON and 360 seconds OFF. However, there still remains a paucity of clinical data on the use of intermittent dosing and which doses (i.e. on/off cycle time periods) are most effective. Furthermore, no previous studies have utilized HF10 therapy when evaluating intermittent dosing.

This study seeks to prospectively compare continuous HF10 therapy versus two intermittent dosing HF10 (ID HF10) therapies - 1) 30 seconds ON and 120 seconds OFF; 2) 30 seconds ON and 360 seconds OFF - in patients endorsing decreasing efficacy of continuous HF10 therapy.

We hypothesize that ID HF10 therapy will provide non-inferior pain relief as measured by NRS scores when compared to continuous HF10 therapy. The primary outcome for this study will be NRS pain scores (0 to 10 where 0 = no pain and 10 = worst pain ever in 0.5 increments). Secondary endpoints include: charging frequency, EQ-5D scores of wellbeing, PROMIS scores for physical function, pain interference, sleep disturbance, and emotional distress; chronic pain acceptance questionnaire 8 (CPAQ-8), patient satisfaction scores, and patient global impression of change.

Patients with chronic back and/or leg pain who have undergone permanent spinal cord stimulator implantation delivered by the Nevro Omnia Neurostimulation System, have had the system in place for at least 1 year, utilizing continuous HF10 therapy, and now endorsing decreasing efficacy of continuous HF10 therapy will be randomized to 2 groups, in a single-blinded, 1:1 fashion:

1. ID HF10 therapy at 30 seconds ON, 90 seconds OFF
2. ID HF10 therapy at 30 seconds ON, 360 seconds OFF

Patient's will be seen and evaluated prior to randomization, and thereafter at 2, 4 and 6 weeks. At the 6-week time period, patients will be crossed over to the other study arm and thereafter evaluated at 2, 4 and 6 weeks.

Randomization will be performed using a computer-generated random sequence generator with equal selection probabilities to all groups. Subjects will be blinded to their randomization.

After randomization, each consented subject will present to clinic at which time will first be seen by a team of investigators, sub-investigators, and/or study staff. After evaluation and collection of baseline data, a clinical specialist for the Nevro Omnia Neurostimulation system will program the subject's SCS system according to the treatment group to which they have been randomized, under direct physician supervision.

Patient will be subsequently seen at 2, 4 and 6-weeks in a clinic setting. At each interval, the patient will be seen by a team of investigators, sub-investigators, and/or study staff to administer questionnaires and collect data. .

Patient specific data to be collected will include:

* Age
* Height
* Weight
* BMI
* Gender
* Primary diagnosis
* Current daily morphine milligram equivalent usage

Data to be collected at baseline and at 6 and 12 weeks of stimulation:

* Patient Health Questionnaire (PHQ-8)
* PROMIS Health questionnaires

  * Global Health 10 item questionnaire
  * Physical Function 8b questionnaire
  * Emotional Distress-8a Anxiety questionnaire
  * Sleep Disturbance 4a questionnaire
  * Fatigue 8 item questionnaire
* CPAQ-8 score (Chronic Pain Acceptance Questionnaire 8)
* Average charging frequency over last week
* Patient Global Impression of Change
* Patient Satisfaction Score

Data to be collected at each study visit:

* NRS pain scores (22-point scale, 0-10 in 0.5 increments)
* Current dorsal root ganglion stimulation parameters (i.e. mode of stimulation-continuous vs. ID, frequency, amplitude, pulse width)
* Average charging frequency over last week (see fig. 1)

Data will be collected and entered on Redcap with data access limited to research personnel. Data will be exported from RedCap™ into an Excel sheets and stored for analysis on the Department of Anesthesiology shared network folder on the Rush domain. Access to this shared resource is limited to research personnel and access is controlled using the users Rush login. The data will be analyzed on an investigators workstation that is password protected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90
* 1-year or more use of continuous HF10 therapy as delivered a permanently implanted Nevro Omnia Neurostimulation System for chronic back and/or leg pain
* Some level of decreasing pain relief from their SCS system (see fig. 3)
* Willing and able to complete protocol requirements, including:

  * Complete health questionnaires and pain scales as specified in the protocol
  * Sign the study-specific informed consent form
  * Complete follow-ups at the designated time periods

Exclusion Criteria:

* Previous intermittent dosing usage and/or failure
* Cervical SCS system
* Other concurrent neuromodulation system in place
* Current daily morphine milligram equivalent usage 90mg or higher

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
NRS pain scores | Up to 3 months
  Subject's Numeric Rating Scale (NRS) score for pain being treated by spinal cord simulation for up to 3 months of designated treatment on a 22 point scale from 0-10 in 0.5 increments with 0 being no pain to 10 being the worse imaginable pain.

SECONDARY OUTCOMES:
Patient Satisfaction with Treatment Score | Up to 3 months
  At each study visit, subjects will rate their satisfaction with their current spinal cord stimulation therapy over the last 3 days as either:
  Completely satisfied, Very satisfied, Slightly Satisfied, Neither satisfied nor dissatisfied, Slightly dissatisfied, Very dissatisfied, Completely dissatisfied
CPAQ-8 | Up to 3 months
  At each study visit, subjects will complete the Chronic Pain Acceptance Questionnaire (CPAQ-8) which asks subjects to rate the truth of different statements about their chronic pain (i.e. I live a full life even though I have chronic pain) as either:
  Never true (0), Very rarely true (1), Seldom true (2), Sometimes true (3), Often true (4), Almost always true (5), Always true (6)
Current mode of stimulation | Up to 3 months
  Spinal cord stimulator settings as either continuous, intermittent dosing 30 seconds ON/120 seconds OFF, or intermittent dosing 30 seconds ON/360 seconds OFF
Stimulator settings- frequency | Up to 3 months
  Subject's current spinal cord stimulator setting frequency in hertz (Hz)
Stimulator settings- amplitude | Up to 3 months
  Subject's current spinal cord stimulator setting amplitude in milliamps (mA)
Stimulator settings- pulse width | Up to 3 months
  Subject's current spinal cord stimulator setting pulse width in microseconds (μs)
Charging frequency of spinal cord stimulator | Up to 3 months
  Average charging frequency over the last week of patient's spinal cord stimulator in hours/minutes.
PROMIS- Fatigue 8 questionnaire | Up to 3 months
  Fatigue 8 questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to feelings of fatigue (i.e. I feel fatigue...) as not at all (1), a little bit (2), somewhat (3), quite a bit (4), or very much (5).
  Subjects will also rate statements pertaining to frequency of fatigue (i.e. How often did you have push yourself to get things done because of your fatigue) as either never (1), rarely (2), sometimes (3), often (4), or always (5).
PROMIS- Sleep Disturbance 4a questionnaire | Up to 3 months
  Sleep Disturbance 4a questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to quality of sleep (i.e. My sleep was refreshing) as either very much (1), quite a bit (2), somewhat (3), a little bit (4), or not at all (5).
  They will also rate their sleep quality as very poor (5), poor (4), fair (3), good (2), or very good (1).
PROMIS- Emotional Distress- 8a Anxiety questionnaire | Up to 3 months
  Emotional Distress- 8a Anxiety questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to feelings of anxiety (i.e. I felt fearful) as either never (1), rarely (2), sometimes (3), often (4), or always (5).
PROMIS- Physical Function 8b questionnaire | Up to 3 months
  Physical Function 8b questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to ability to do physical tasks (i.e. Are you able to run errands and shop) as either unable to do (1), with much difficulty (2), with some difficulty(3), with a little difficulty (4), or without any difficulty (5).
  They will also rate statements pertaining to any health limitations on physical functions (i.e. Does your health now limit you in lifting or carrying groceries) as not at all (5), very little (4), somewhat (3), quite a lot (2), or cannot do (1).
PROMIS- Pain Interference 6b questionnaire | Up to 3 months
  Pain Interference 6b questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining the extent that pain interferes with their life (i.e. How much did pain interfere with your enjoyment of life) as either not at all (1), a little bit (2), somewhat (3), quite a bit (4), or very much (5).
  They will answer how much pain kept them from socializing with others in the past 7 days as either never (5), rarely (4), sometimes (3), often (2), or always (1).
PROMIS- Global Health 10 item questionnaire | Up to 3 months
  Global Health 10 item questionnaire outcome at up to 3 months on designated treatment. Subjects will rate statements pertaining to their overall health (i.e. In general, would you say your quality of life is) as either poor (1), fair(2), good (3), very good (4), or excellent (5).
PHQ-8 | Up to 3 months
  At each study visit, subjects will complete the Patient Health Questionnaire (PHQ-8) which asks subjects to rate over the past 2 weeks how often they feel a particular emotion (i.e. feeling tired or having little energy) as either
  Not at all, Several days, More than half the days, Nearly every day
  If any problems were checked off, subjects will rate how difficult these problems made it to do work, take care of things at home, or get along with others as either:
  Not difficult at all, Somewhat difficult, Very difficult, Extremely difficult
Patient Global Impression of Change | Up to 3 months
  At each study visit, subjects will be asked to rate their progress with the current spinal cord stimulator therapy over the last 3 days compared to their paresthesia SCS therapy as either:
  Very much improved, Much improved, Minimally improved, No change, Minimally worse, Much worse, Very much worse

CONTACTS AND LOCATIONS:
Overall Officials: Robert J McCarthy, PharmD, Study Director — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No
Available upon reasonable request from principal investigator.

REFERENCES:
- [Background] Kapural L, Yu C, Doust MW, Gliner BE, Vallejo R, Sitzman BT, Amirdelfan K, Morgan DM, Brown LL, Yearwood TL, Bundschu R, Burton AW, Yang T, Benyamin R, Burgher AH. Novel 10-kHz High-frequency Therapy (HF10 Therapy) Is Superior to Traditional Low-frequency Spinal Cord Stimulation for the Treatment of Chronic Back and Leg Pain: The SENZA-RCT Randomized Controlled Trial. Anesthesiology. 2015 Oct;123(4):851-60. doi: 10.1097/ALN.0000000000000774. PMID 26218762
- [Background] Miller JP, Eldabe S, Buchser E, Johanek LM, Guan Y, Linderoth B. Parameters of Spinal Cord Stimulation and Their Role in Electrical Charge Delivery: A Review. Neuromodulation. 2016 Jun;19(4):373-84. doi: 10.1111/ner.12438. Epub 2016 May 6. PMID 27150431
- [Background] Deer T, Slavin KV, Amirdelfan K, North RB, Burton AW, Yearwood TL, Tavel E, Staats P, Falowski S, Pope J, Justiz R, Fabi AY, Taghva A, Paicius R, Houden T, Wilson D. Success Using Neuromodulation With BURST (SUNBURST) Study: Results From a Prospective, Randomized Controlled Trial Using a Novel Burst Waveform. Neuromodulation. 2018 Jan;21(1):56-66. doi: 10.1111/ner.12698. Epub 2017 Sep 29. PMID 28961366
- [Background] Alo KM, Redko V, Charnov J. Four Year Follow-up of Dual Electrode Spinal Cord Stimulation for Chronic Pain. Neuromodulation. 2002 Apr;5(2):79-88. doi: 10.1046/j.1525-1403.2002.02017.x. PMID 22151846
- [Background] Turner JA, Loeser JD, Deyo RA, Sanders SB. Spinal cord stimulation for patients with failed back surgery syndrome or complex regional pain syndrome: a systematic review of effectiveness and complications. Pain. 2004 Mar;108(1-2):137-47. doi: 10.1016/j.pain.2003.12.016. PMID 15109517
- [Background] Hayek SM, Veizi E, Hanes M. Treatment-Limiting Complications of Percutaneous Spinal Cord Stimulator Implants: A Review of Eight Years of Experience From an Academic Center Database. Neuromodulation. 2015 Oct;18(7):603-8; discussion 608-9. doi: 10.1111/ner.12312. Epub 2015 Jun 5. PMID 26053499
- [Background] Pope JE, Deer TR, Falowski S, Provenzano D, Hanes M, Hayek SM, Amrani J, Carlson J, Skaribas I, Parchuri K, McRoberts WP, Bolash R, Haider N, Hamza M, Amirdelfan K, Graham S, Hunter C, Lee E, Li S, Yang M, Campos L, Costandi S, Levy R, Mekhail N. Multicenter Retrospective Study of Neurostimulation With Exit of Therapy by Explant. Neuromodulation. 2017 Aug;20(6):543-552. doi: 10.1111/ner.12634. Epub 2017 Jul 17. PMID 28714533
- [Background] Van Buyten JP, Wille F, Smet I, Wensing C, Breel J, Karst E, Devos M, Poggel-Kramer K, Vesper J. Therapy-Related Explants After Spinal Cord Stimulation: Results of an International Retrospective Chart Review Study. Neuromodulation. 2017 Oct;20(7):642-649. doi: 10.1111/ner.12642. Epub 2017 Aug 18. PMID 28834092
- [Background] Vesper J, Slotty P, Schu S, Poeggel-Kraemer K, Littges H, Van Looy P, Agnesi F, Venkatesan L, Van Havenbergh T. Burst SCS Microdosing Is as Efficacious as Standard Burst SCS in Treating Chronic Back and Leg Pain: Results From a Randomized Controlled Trial. Neuromodulation. 2019 Feb;22(2):190-193. doi: 10.1111/ner.12883. Epub 2018 Nov 19. PMID 30456795
- [Background] Deer TR, Patterson DG, Baksh J, Pope JE, Mehta P, Raza A, Agnesi F, Chakravarthy KV. Novel Intermittent Dosing Burst Paradigm in Spinal Cord Stimulation. Neuromodulation. 2021 Apr;24(3):566-573. doi: 10.1111/ner.13143. Epub 2020 Mar 23. PMID 32202044